CLINICAL TRIAL: NCT04088331
Title: Artificial Urinary Sphincter Clinical Outcomes
Acronym: AUSCO
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: U0669
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Results first posted 2025-08-03 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AMS 800 Artificial Urinary Sphincter Recipients: Adult males with moderate to severe primary stress urinary incontinence (as assessed by a baseline pad weight test) due to ISD who meet the indications for surgical correction of urinary incontinence.
  Interventions: Device: AMS 800 Artificial Urinary Sphincter

INTERVENTIONS:
Device: AMS 800 Artificial Urinary Sphincter — The AMS 800 Artificial Urinary Sphincter (AUS) is an implantable, fluid filled, solid silicone elastomer device used to treat stress urinary incontinence due to reduced urethral/bladder outlet resistance (intrinsic sphincter deficiency). It is designed to restore the natural process of urinary control. The device simulates normal sphincter function by opening and closing the urethra under the control of the patient.

SUMMARY:
To evaluate the AMS 800 Artificial Urinary Sphincter (AUS) in men with primary stress urinary incontinence as measured by pad weight tests.

DETAILED DESCRIPTION:
Study is designed to evaluate the performance of the AMS 800 Artificial Urinary Sphincter (AUS) in men with primary stress urinary incontinence as measured by pad weight tests.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. ≥ 18 years of age
3. Has undergone either a radical prostatectomy, transurethral resection of the prostate or other invasive prostate surgery
4. Demonstrates primary stress urinary incontinence
5. Positive screening 24-hour pad weight test (≥100 grams)
6. Experiences at least 3 incontinence episodes per day during baseline diary or presents with continuous incontinence
7. Negative urine culture
8. Willing and able to undergo surgical implantation of the AUS device
9. Willing and able to comply with the follow-up requirements
10. Willing and able to forego any other surgical urinary incontinence treatments while participating in the study
11. Willing and able to sign the informed consent

Exclusion Criteria:

1. Previously had or currently has a device implanted (AUS/Sling, or otherwise) for treatment of SUI or urge incontinence
2. Primary urgency incontinence
3. Postvoid residual volume greater that 150 ml or a history of difficulty emptying the bladder
4. Recurrent vesicourethral anastomotic stricture or urethral stricture disease within the past 6 months
5. Known urogenital malignancy other than previously treated prostate cancer
6. Recurrent prostate cancer that is expected to require intervention during the study follow-up period
7. History of recurrent bladder stones within the past 12 months prior to signing the informed consent
8. Neurogenic bladder
9. Need for intermittent catheterization
10. Known history of bleeding diathesis or coagulopathy
11. Immunosuppressed or on medical therapy which would impact the immune system
12. Uncontrolled diabetes, defined as (HbA1c>10)
13. Has a genitourinary mechanical prosthesis that was implanted within 3 months from the date of consent
14. Had a post-implantation infection associated with the device after genitourinary mechanical prosthesis was implanted
15. Undergone bulking procedure within 6 months of the baseline assessment
16. Poor candidate for surgical procedures and/or anesthesia due to physical or mental conditions
17. Urinary incontinence due to or complicated by an irreversibly obstructed lower urinary tract
18. Irresolvable detrusor hyperreflexia or bladder instability
19. Currently enrolled or plans to enroll in another device or drug clinical trial
20. Currently using an indwelling catheter or condom catheter for treatment of incontinence and is not willing to discontinue use at least 4 weeks prior to baseline assessment
21. Known allergy or sensitivity to rifampin or to minocycline HCl or other tetracyclines (only applicable when implanting with InhibiZone version of this device)
22. Systemic lupus erythematosus because minocycline HCl has been reported to aggravate this condition (only applicable when implanting with InhibiZone version of this device)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll adult males with moderate to severe primary stress urinary incontinence (as assessed by a baseline pad weight test) due to ISD who meet the indications for surgical correction of urinary incontinence.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Kaufman, MD, Principal Investigator — Vanderbilt Urology
Locations (18):
- United States (16):
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Hospital, Aurora, Colorado
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - Willis-Knighton Bossier Medical Center, Bossier City, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Lahey Clinic Hospital, Burlington, Massachusetts
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - Urology San Antonio Research, PA., San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
- Australia (2):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Australian Urology Associates, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaufman MR, Wood HM, Terlecki R, Moon D, Myers J, Vanni AJ, Jones L, Broghammer JA, Henry G, Breyer BN, Erickson B, Burnett AL, Johnsen NV, Loong Chan LW, Flynn BJ, Khavari R, Smith TG 3rd, Elliott S, Chaussee EL, Rainbow K, Peterson AC. The Artificial Urinary Sphincter Clinical Outcomes Trial: Primary Results. J Urol. 2026 Feb;215(2):194-202. doi: 10.1097/JU.0000000000004796. Epub 2025 Oct 3. PMID 41042705

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects will be considered enrolled in the study once they sign the informed consent. All enrolled subjects will have been consented prior to the procedure. All enrolled subjects with a surgery initiated (i.e. first incision) will be considered part of the Intent-to-Treat (ITT) population. A total of 145 subjects were enrolled and 115 continued on to undergo the index procedure, qualifying them for inclusion in the ITT population.
Period: Overall Study
Arm/Group | AMS 800 Artificial Urinary Sphincter Recipients
Started | 115
Completed | 101
Not Completed | 14
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 7
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Arm/Group | AMS 800 Artificial Urinary Sphincter Recipients
Number analyzed (Participants) | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 98
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 115
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 100
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 109
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Reduction in 24 Hour Pad Weight Test at 12 Months
Description: Number of subjects achieving 50% reduction or greater in baseline urinary incontinence as measured by 24-hour pad weight test at 12 months post device activation
Time Frame: 12 months
Population: The analysis was performed on subjects in the Intent to Treat (ITT) population who had available 24-hr pad weight data available at their 12 month follow-up visit. The ITT subject population included all subjects who provided written informed consent to be enrolled into the study, and have a surgery initiated (defined as the first incision).
Measure: Count of Participants; unit: Participants
Arm/Group | AMS 800 Artificial Urinary Sphincter Recipients
Number analyzed (Participants) | 97
Participants | 91
Statistical Analysis 1: Comparison: AMS 800 Artificial Urinary Sphincter Recipients; Hypotheses: H0: p ≤ 0.65 H1: p > 0.65 where p = the proportion of subjects who are a treatment success. Hypotheses evaluated using a one-sided exact binomial test. Power calculation assumed a treatment success rate of 80%. With a one-sided type I error of 0.025 and a type II error of 0.10 (90% power), a sample size of 96 subjects needed to demonstrate the proportion of subjects who are a treatment success exceeds 65%; Test type: Superiority; p < 0.001, Exact binomial test

2. Secondary Outcome: Percentage of Participants That Required Revision (Revision Rates), Had Serious Adverse Events, and Had Serious Adverse Events That Are Device and/or Procedure Related
Description: Percentage of Participants that Required Revision (Revision Rates), had Serious Adverse Events, and had Serious Adverse Events that are Device and/or Procedure Related at 3 months, 6 months, and 12 months. Adverse event and revision rates are summarized by the Kaplan-Meier estimate with revision/event timing relative to the index procedure.
Time Frame: 3 months, 6 months, and 12 months
Population: The analysis was performed for the Intent to Treat (ITT) population. The ITT subject population included all subjects who provided written informed consent to be enrolled into the study, and have a surgery initiated (defined as the first incision).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | AMS 800 Artificial Urinary Sphincter Recipients
Number analyzed (Participants) | 115
Percentage of participants
  Incidence of Safety Parameters at 3 months: Revision Rates | 3.5 [1.3 to 9.1]
  Incidence of Safety Parameters at 3 months: Serious adverse events | 9.6 [5.5 to 16.7]
  Incidence of Safety Parameters at 3 months: SAEs that are device and/or procedure related | 5.2 [2.4 to 11.3]
  ncidence of Safety Parameters at 6 months: Revision Rates | 6.2 [3.0 to 12.6]
  Incidence of Safety Parameters at 6 months: Serious adverse events | 12.4 [7.5 to 20]
  Incidence of Safety Parameters at 6 months: SAEs that are device and/or procedure related | 7.0 [3.6 to 13.6]
  Incidence of Safety Parameters at 12 months: Revision Rates | 7.2 [3.7 to 13.8]
  Incidence of Safety Parameters at 12 months: Serious adverse events | 15.2 [9.7 to 23.3]
  Incidence of Safety Parameters at 12 months: SAEs that are device and/or procedure related | 8.9 [4.9 to 16.0]

3. Secondary Outcome: Number of Subjects Achieving ≥ 50% Reduction in 24 Hour Pad Weight Test at Device Activation
Description: Number of subjects achieving ≥ 50% reduction in urinary incontinence as measured by 24-hour pad weight test at device activation compared to baseline
Time Frame: Device Activation
Population: 107 subjects had data at both baseline and device activation.
Measure: Count of Participants; unit: Participants
Arm/Group | AMS 800 Artificial Urinary Sphincter Recipients
Number analyzed (Participants) | 107
Participants | 75

4. Secondary Outcome: Number of Subjects Achieving ≥ 75% Reduction in 24 Hour Pad Weight Test at Device Activation
Description: ≥ 75% reduction in urinary incontinence as measured by 24-hour pad weight test at device activation compared to baseline
Time Frame: Device Activation
Measure: Count of Participants; unit: Participants
Arm/Group | AMS 800 Artificial Urinary Sphincter Recipients
Number analyzed (Participants) | 107
Participants | 70

5. Secondary Outcome: Change in Number of Pads Per Day at 3 Months
Description: Change in number of pads per day at 3 months compared to baseline. Change was calculated by subtracting the number of pads per day at baseline from the number of pads per day at 3 months.
Time Frame: 3 months
Population: 109 subjects had data at both baseline and 3 months post device activation.
Measure: Mean (95% Confidence Interval); unit: Pads per day
Arm/Group | AMS 800 Artificial Urinary Sphincter Recipients
Number analyzed (Participants) | 109
Pads per day | -4.0 [-4.4 to -3.5]

6. Secondary Outcome: Number of Subjects Achieving ≥ 50% Reduction in 24 Hour Pad Weight Test at 6 Months
Description: Number of subjects achieving ≥ 50% reduction in urinary incontinence as measured by 24-hour pad weight test at 6 months post device activation compared to baseline
Time Frame: 6 months
Population: 99 subjects had data at both baseline and 6 months post device activation.
Measure: Count of Participants; unit: Participants
Arm/Group | AMS 800 Artificial Urinary Sphincter Recipients
Number analyzed (Participants) | 99
Participants | 88

7. Secondary Outcome: Number of Subjects Achieving ≥ 75% Reduction in 24 Hour Pad Weight Test at 6 Months
Description: ≥ 75% reduction in urinary incontinence as measured by 24-hour pad weight test at 6 months post device activation compared to baseline
Time Frame: 6 months
Population: 99 subjects had data at both baseline and 6 months post device activation.
Measure: Count of Participants; unit: Participants
Arm/Group | AMS 800 Artificial Urinary Sphincter Recipients
Number analyzed (Participants) | 99
Participants | 84

8. Secondary Outcome: Number of Subjects Achieving ≥ 75% Reduction in 24 Hour Pad Weight Test at 12 Months
Description: ≥ 75% reduction in urinary incontinence as measured by 24-hour pad weight test at 12 months post device activation compared to baseline
Time Frame: 12 months
Population: 97 subjects had data at both baseline and 6 months post device activation.
Measure: Count of Participants; unit: Participants
Arm/Group | AMS 800 Artificial Urinary Sphincter Recipients
Number analyzed (Participants) | 97
Participants | 83

9. Secondary Outcome: Change in Number of Pads Per Day at 6 Months
Description: Change in number of pads per day at 6 months post-device activation compared to baseline. Change was calculated by subtracting the number of pads per day at baseline from the number of pads per day at 6 months.
Time Frame: 6 months
Population: 99 subjects had data at both baseline and 6 months post device activation.
Measure: Mean (95% Confidence Interval); unit: Pads per day
Arm/Group | AMS 800 Artificial Urinary Sphincter Recipients
Number analyzed (Participants) | 99
Pads per day | -4.0 [-4.5 to -3.5]

10. Secondary Outcome: Change in Number of Pads Per Day at 12 Months
Description: Change in number of pads per day at 12 months post-device activation compared to baseline. Change was calculated by subtracting the number of pads per day at baseline from the number of pads per day at 12 months.
Time Frame: 12 months
Population: 101 subjects had data at both baseline and 12 months post device activation.
Measure: Mean (95% Confidence Interval); unit: Pads per day
Arm/Group | AMS 800 Artificial Urinary Sphincter Recipients
Number analyzed (Participants) | 101
Pads per day | -3.9 [-4.4 to -3.4]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of index procedure through study completion, which was up to 12 months post-device activation.
Description: AE reporting included: Serious Adverse Events, Serious Adverse Device Effects, Adverse Device Effects, and Procedure Related Adverse Events
Arm/Group | AMS 800 Artificial Urinary Sphincter Recipients
All-Cause Mortality (participants affected / at risk) | 3/115
Serious Adverse Events (participants affected / at risk) | 17/115
Other Adverse Events (participants affected / at risk) | 27/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMS 800 Artificial Urinary Sphincter Recipients (N=115)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Death (General disorders) | 1 (1)
Medical device site erosion (General disorders) | 1 (1)
Medical device site induration (General disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1)
Labyrinthitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Device dislocation (Product Issues) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Incontinence (Renal and urinary disorders) | 1 (1)
Renal mass (Renal and urinary disorders) | 1 (1)
Urinary fistula (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urothelium erosion (Renal and urinary disorders) | 1 (1)
Medical device change (Surgical and medical procedures) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMS 800 Artificial Urinary Sphincter Recipients (N=115)
Localized oedema (General disorders) | 1 (1)
Medical device site discomfort (General disorders) | 2 (2)
Medical device site haematoma (General disorders) | 1 (1)
Medical device site reaction (General disorders) | 1 (1)
Postoperative wound infection (Infections and infestations) | 3 (3)
Scrotal infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1)
Incision site swelling (Injury, poisoning and procedural complications) | 1 (1)
Scrotal haematoma (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Pudendal canal syndrome (Nervous system disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1)
Urethritis noninfective (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 3 (3)
Oedema genital (Reproductive system and breast disorders) | 1 (1)
Perineal pain (Reproductive system and breast disorders) | 1 (1)
Scrotal erythema (Reproductive system and breast disorders) | 1 (1)
Scrotal swelling (Reproductive system and breast disorders) | 3 (3)
Testicular pain (Reproductive system and breast disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT04088331/Prot_SAP_000.pdf